CLINICAL TRIAL: NCT06974825
Title: A Randomized, Double-blind, Placebo and Positive Drug Parallel-controlled Phase IIa Clinical Study Protocol to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Characteristics of Multiple-dose BGM0504 Injection in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of BGM0504 in Chinese Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BrightGene Bio-Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BGM0504-IIa-T2DM
Record Dates: First submitted 2025-05-14; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 5 mg BGM0504 (Experimental)
  Interventions: Drug: BGM0504 Administered SC
- 10 mg BGM0504 (Experimental)
  Interventions: Drug: BGM0504 Administered SC
- 15 mg BGM0504 (Experimental)
  Interventions: Drug: BGM0504 Administered SC
- 1 mg Semaglutide (Experimental)
  Interventions: Drug: Semaglutide Administered SC
- Placebo (Experimental)
  Interventions: Drug: Placebo Administered SC

INTERVENTIONS:
Drug: BGM0504 Administered SC — 5 milligrams (mg) BGM0504 administered subcutaneously (SC) once a week.
  Arms: 5 mg BGM0504
Drug: BGM0504 Administered SC — Experimental: 10 mg BGM0504 10 mg BGM0504 administered SC once a week.
  Arms: 10 mg BGM0504
Drug: BGM0504 Administered SC — Experimental: 15 mg BGM0504 15 mg BGM0504 administered SC once a week.
  Arms: 15 mg BGM0504
Drug: Semaglutide Administered SC — Active Comparator: 1 mg Semaglutide
  1 mg semaglutide administered SC once a week
  Arms: 1 mg Semaglutide
Drug: Placebo Administered SC — Placebo Comparator: Placebo Placebo administered SC once a week.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of BGM0504 in Chinese patients with Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with type 2 diabetes mellitus (T2DM);
* Glycosylated hemoglobin (HbA1c) at screening/baseline: 7.0% ≤ HbA1c ≤ 10%;
* Body Mass Index (BMI): 19.5 kg/m2 ≤ BMI ≤ 35.0 kg/m2;
* Fasting blood glucose (FPG) at screening/baseline: FPG ≤ 13.3 mmoL/L

Exclusion Criteria:

* Diagnosed with non-type 2 diabetes mellitus;
* Grade 3 hypoglycemia within 6 months prior to screening;
* Concomitant thyroid dysfunction that cannot be controlled at a stable drug dose at screening, or clinically significant abnormalities in thyroid function test results at screening that require initiation of therapy;
* Subjects with uncontrolled hypertension after treatment (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg at screening) or untreated blood pressure meeting the above criteria at screening;
* Patients with a previous history or clinical evidence of acute or chronic pancreatitis;
* Malignant tumor confirmed within 5 years prior to screening (except cured carcinoma in situ) or potential malignant tumor assessed at screening;
* Patients with severe mental illness or language disorder at screening, unwilling or unable to fully understand and cooperate;
* Female subjects during pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Hemoglobin A1c (HbA1c) | Week 0 to Week 12
  Change from baseline in HbA1c after 12 weeks of treatment.

SECONDARY OUTCOMES:
Change From Baseline in Body Weight | Week 0 to Week 12
  Change from baseline in body weight after 12 weeks of treatment.
Percentage of Participants With HbA1c Target Value of <7% | Week 0 to Week 12
  Percentage of Participants With HbA1c Target Value of <7% after 12 weeks of treatment.
Percentage of Participants With HbA1c Target Value of <6.5% | Week 0 to Week 12
  Percentage of Participants With HbA1c Target Value of <5.7% after 12 weeks of treatment.
Change From Baseline in Fasting Serum Glucose | Week 0 to Week 12
  Change from baseline in FPG after 12 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China